CLINICAL TRIAL: NCT07090629
Title: The Benefits of the Measureof Epicardial Adipose Tissue During Coronary Calcium Assessment of the Refine Cardiovascular Risk Assessment at Reunion Island.
Acronym: EPICAC-RUN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Aix Marseille Université (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/CHU/21; 2024/CHU/21 (Other: CHU de La Réunion)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: High Cholesterol; Lipodystrophy, Familial Partial; Diabetes
Keywords: coronary calcium score; epicardial adipose tissue; cardiovascular risk scoring; lipodystrophy
MeSH Terms: conditions — Hypercholesterolemia; Lipodystrophy, Familial Partial; Diabetes Mellitus; Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Partial Lipodystrophy, Type 2 (FPLD): Adult patients with a confirmed genetic diagnosis of lipodystrophy
  Interventions: Other: Epicardial adipose tissue measurement on the available tododensitometry used for coronary calcium scoring
- Control group of patients at high cardiovascular risk (CTL): Patients without Familial Partial Lipodystrophy
  Interventions: Other: Epicardial adipose tissue measurement on the available tododensitometry used for coronary calcium scoring

INTERVENTIONS:
Other: Epicardial adipose tissue measurement on the available tododensitometry used for coronary calcium scoring — Epicardial adipose tissue measurement

SUMMARY:
The goal of this retrospective study is to see whether patients with familial partial type 2 lipodystrophy, who are at high cardiovascular risk present a higher volume of visceral epicardial adipose tissue than other patients without familial partial lipodystrophy who were assessed for their cardiovascular risk using coronary artery calcification scoring between 2016 and 2024.

DETAILED DESCRIPTION:
Coronary artery calcification and clinical cardiovascular risk scoring are insufficient for patients with Familial Partial Lipodystrophy Part 2 (FPLD2), who often develop cardiovascular events before 40 and are insulin resistant. Epicardial adipose tissue volume could be a new, earlier marker of interest for these patients related to inflammation and atherosclerosis. The investigators retrospectively included high cardiovascular risk patients from 2016 to 2023 who had benefited from coronary artery calcification and clinical risk scoring at the University Hospital of La Réunion with Familial Partial Lipodystrophy Type 2 or controls and paired them for age, sex and body mass index. Epicardial adipose tissue volume was measured on the same tododensitometry as the CAC scoring, using a semi, automated technique that had been validated with deep learning at the Univeristy Hospital of Aix-Marseille.

ELIGIBILITY:
Inclusion Criteria:

Patients who received a check-up for hypercholesterolemia, obesity or diabetes including a CT scan to measure the coronary calcium score at the CHU de La Réunion between 2016 and 2023

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a check-up for hypercholesterolemia, obesity or diabetes including a CT scan to measure the coronary calcium score at the CHU de La Réunion between 2016 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Epicardial adipose tissue volume | at inclusion
  in mL

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No